CLINICAL TRIAL: NCT05884034
Title: Effects of a Self-care Educational Program Via Telerehabilitation on Quality of Life and Caregiver Burden in Amyotrophic Lateral Sclerosis: Randomized Clinical Trial Protocol
Brief Title: Effects of a Self-care Educational Program Via Telerehabilitation in Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Ana Raquel Rodrigues Lindquist, PhD, Research group leader, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CEP/UFRN 4.076.825/20
Record Dates: First submitted 2023-05-18; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Quality of Life
Keywords: Caregiver; Caregiver Burden; Telemedicine
MeSH Terms: conditions — Caregiver Burden | interventions — Telerehabilitation; Educational Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): Self-care educational program via telerehabilitation
  Interventions: Other: Telerehabilitation
- Education group (Active Comparator): Self-care educational program via informative booklet
  Interventions: Other: Education

INTERVENTIONS:
Other: Telerehabilitation — Subjects will participate in a six-week self-care education program with weekly synchronous meetings using Google Meet or WhatsApp and an informative booklet containing guidelines for performing physical activities at home and information on healthy eating, mental health and routine management, with a schedule for weekly organization.
  Arms: Telerehabilitation group
Other: Education — Participants will receive an informative booklet containing guidelines for performing physical activities at home and information on healthy eating, mental health and routine management, with orientations on the importance of reading and implementing the guidelines described in the booklet.
  Arms: Education group

SUMMARY:
The purpose of this study is to evaluate the effects of a self-care educational program via telerehabilitation on the quality of life, burden, stress, pain, and depression of caregivers of people with ALS.

DETAILED DESCRIPTION:
This study is a randomized clinical trial that will be developed at the Laboratory of Intervention and Analysis of Movement (LIAM) of the Physiotherapy Department of the Federal University of Rio Grande do Norte (UFRN). The participants of this study will comprise informal caregivers of ALS people living in the municipalities of Natal (Rio Grande do Norte, Brazil), aged 18 years or above, of both sexes. The research sample will be allocated randomly into two distinct groups: control group (GC) and experimental group (GE). This research was submitted to the Research Ethics Committee (REC) (no. 4.076.825/20). All participants will be informed about the aim of the study before the program and sign the informed consent form, following the Resolution 466/2012 of the National Health Council and the Declaration of Helsinki.

All participants will undergo an assessment at baseline, immediately after the six-week program, and 30 days after the end of the program. A researcher not involved in the intervention will conduct all evaluations remotely via Whatsapp or Google Meet. Analyzed outcomes include the caregiver burden (Zarit scale), quality of life (World Health Organization Quality of Life Bref), pain (McGill Pain Questionnaire), stress (Perceived Stress Scale), and depression (Beck Depression Inventory).

GE group will receive an informative booklet for caregivers in person and will be divided into subgroups. Each subgroup will participate in a six-week self-care education program with weekly synchronous meetings using Google Meet or WhatsApp. Each meeting will address topics related to the physical and mental health of caregivers, including the importance of care and caregivers, physical activities to be performed at home, routine management and healthy eating.

Participants allocated to the CG group will receive the same booklet. In addition, they will receive guidance on the importance of reading and applying the guidelines in the booklet. After the baseline assessment, trained researchers will contact the participants in the second and sixth week of the study to verify their physical and mental health and whether they are performing physical activities and having difficulties living with the individual with ALS.

ELIGIBILITY:
Inclusion Criteria:

* Informal caregiver (i.e., family member, friend, or a caregiver without payment) of an individual with ALS (clinically defined, probable, or possible) diagnosed by a neurologist using the (El Escorial Criteria);
* Informal caregiver of people who did not have any other neurological disease associated with ALS;
* Aged 18 years or above;
* Without cognitive impairment on the Mini-Mental State Examination (MMSE; cutoff point of 25 for literate individuals) for understanding the study and the informed consent form;
* Literate (at least complete primary education).

Exclusion Criteria:

* Health conditions that hinder from exercising safely, such as recent surgeries, fractures; uncontrolled heart, vascular and respiratory disorders; dizziness or vertigo, fainting; oncological diseases; neurological diseases that affect balance and protective reactions;
* Caregivers in the first trimester of pregnancy, due to the risk of the sudden increase in resting heart rate;
* Using psychiatric medication, such as anxiolytics, antidepressants, antipsychotics, and antiepileptics, as the use of these medications may interfere with the results of this study;
* Drop out of two or more consecutive days without replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in caregiver burden score measured through Zarit scale | Baseline, immediately after the intervention protocol, and after 4 weeks after treatment
  Measured through Zarit scale. The analyzed variable will be the score obtained from 22 questions scored on a 5-point Likert scale, from 0 (never) to 4 (nearly always)

SECONDARY OUTCOMES:
Change in quality of life score measured through World Health Organization Quality of Life-100 (WHOQOL-BREF) | Baseline, immediately after the intervention protocol, and after 4 weeks after treatment
  Measured through World Health Organization Quality of Life-100 (WHOQOL) BREF, wich is a 0-100 scale scored in a positive direction (i.e. higher scores denote higher quality of life). The analyzed variable will be the score obtained from 26 questions.
Change in pain score measured through McGill Pain Questionnaire | Baseline, immediately after the intervention protocol, and after 4 weeks after treatment
  Measured through McGill Pain Questionnaire, wich is a 0-78 scale scored in a negative direction (i.e. higher scores denote higher pain). The analyzed variable will be the score obtained from 78 descriptors of pain organized into four categories (sensory, affective, evaluative, and miscellaneous) and 20 subcategories.
Change in stress score measured through Perceived Stress Scale (PSS) | Baseline, immediately after the intervention protocol, and after 4 weeks after treatment
  Measured through PSS. The analyzed variable will be the score obtained from 14 questions scoring from 0 to 4 (0 = never, 1 = almost never, 2 = sometimes, 3 = almost always, and 4 = always).
Change in depressive symptoms evaluated through Beck Depression Inventory | Baseline, immediately after the intervention protocol, and after 4 weeks after treatment
  Measured through Beck Depression Inventory, wich is a 0-63 scale scored in a negative direction (i.e. higher scores denote more depression). The analyzed variable will be the score obtained from 21 items regarding attitudes and symptoms of depression.
Change in night awakenings measured through Sênior Saúde Móvel platform | Baseline, daily during the entire intervention protocol, and after 4 weeks after treatment
  Measured by Sênior Saúde Móvel platform. This data will be acquired through a wearable device and used in specific applications of algorithms capable of performing the screening and will be automatically sent to the Sênior Saúde Móvel platform.
Change in sleep patterns measured through Sênior Saúde Móvel platform | Baseline, daily during the entire intervention protocol, and after 4 weeks after treatment
  Measured by Sênior Saúde Móvel platform.
Change in level of physical activity measured through Sênior Saúde Móvel platform | Baseline, daily during the entire intervention protocol, and after 4 weeks after treatment
  Measured by Sênior Saúde Móvel platform.
Change in heart rate variability measured through Sênior Saúde Móvel platform | Baseline, daily during the entire intervention protocol, and after 4 weeks after treatment
  Measured by Sênior Saúde Móvel platform.

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Lindquist, PhD, Study Chair — Universidade Federal do Rio Grande do Norte
Locations (1):
- Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

REFERENCES:
- [Derived] Gomes de Souza E Silva EM, Tomaz da Silva S, Januario de Holanda L, Tezoni Borges D, Mendonca Fernandes AP, Evangelista Rodrigues da Silva K, Souza Ribeiro T, Protasio de Melo L, de Medeiros Valentim RA, Alves Pinto Nagem D, Rodrigues Lindquist AR. Effects of a self-care educational program via telerehabilitation on quality of life and caregiver burden in amyotrophic lateral sclerosis: a single-blinded randomized clinical trial protocol. Front Psychol. 2023 Aug 17;14:1164370. doi: 10.3389/fpsyg.2023.1164370. eCollection 2023. PMID 37663359